CLINICAL TRIAL: NCT01910155
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Design, Multiple-Site Study to Evaluate the Clinical Equivalence of Ciprofloxacin 0.3%/Dexamethasone 0.1% Sterile Otic Suspension (Par) Compared to CIPRODEX® (Ciprofloxacin 0.3%/Dexamethasone 0.1%) Sterile Otic Suspension (Alcon) in the Treatment of Adults With Acute Bacterial Otitis Externa
Brief Title: A Bioequivalence Study of Two Ciprofloxacin/Dexamethasone Formulations in Patients With Otitis Externa
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: FDA's draft guidance (March 2015) provided option of in-vitro or in-vivo studies for bioequivalence. Small study size resulted in negative culture rates.
Sponsor: Par Pharmaceutical, Inc. (Industry)
Collaborators: Novum Pharmaceutical Research Services (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 71205502
Record Dates: First submitted 2013-07-25; First posted 2013-07-29 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Otitis Externa
MeSH Terms: conditions — Otitis Externa | interventions — Ciprofloxacin; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test (Experimental): Ciprofloxacin/Dexamethasone
  Interventions: Drug: Ciprofloxacin/Dexamethasone
- Reference (Active Comparator): Ciprodex (R)
  Interventions: Drug: Ciprodex (R)
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciprofloxacin/Dexamethasone
  Arms: Test
Drug: Ciprodex (R)
  Arms: Reference
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of this study is to compare the relative efficacy and safety of the test formulation of ciprofloxacin 0.3%/dexamethasone 0.1% sterile otic suspension (Par Pharmaceutical Companies, Inc.) to the already-marketed formulation CIPRODEX® (ciprofloxacin 0.3%/dexamethasone 0.1%) sterile otic suspension (Alcon) in the treatment of acute bacterial otitis externa.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non lactating females 18-65 years of age inclusive.
2. Signed informed consent form, which meets all of the criteria of current FDA regulations.
3. If female and of child bearing potential, have a negative urine pregnancy test at the baseline visit and prepare to abstain from sexual intercourse or use a reliable method of contraception during the study (e.g., condom, IUD, oral, injected, transdermal or implanted hormonal contraceptives). Patients on hormonal contraceptives must have been on the same method/type for at least 28 days prior to the start of the study and remain on the same throughout the study.
4. The presence of infection confirmed by a positive bacterial culture for the presence of Pseudomonas aeruginosa or Staphylococcus aureus. As the results of the bacterial culture will not be immediately known, patients who meet all the other inclusion/exclusion criteria may be enrolled in the study pending the results of the bacterial culture.
5. Clinical signs and symptoms consistent with bacterial otitis externa as defined by a combined Total Symptom Score (TSS) of at least 6 with a score of least 2 for otalgia using the following scale 0=none, 1=mild, 2=moderate, 3=severe.

Exclusion Criteria:

1. Females who are pregnant, breast feeding, or anticipate becoming pregnant during the study.
2. Signs and symptoms of otitis externa for longer than 21 days prior to being screened for inclusion in the study.
3. Previous episode of otitis externa within the previous 6 months or more than 2 episodes within the previous 12 months.
4. Been provided any therapeutic drug treatment for current episode of otitis externa.
5. Known history of, or ear exam reveals tympanic membrane perforation or damage for any reason.
6. Current or previous history of any otologic surgery including insertion/removal of tympanostomy tubes in infected ear(s).
7. Clinical diagnosis that suggests current signs or symptoms are not caused by acute bacterial otitis externa e.g. chronic suppurative otitis externa, acute otitis media
8. Clinical diagnosis of malignant otitis externa
9. Mastoid cavities, stenosis, exostosis or tumors of either ear or other noninfectious diseases of either ear.
10. Suspected concurrent fungal or viral infection (e.g. herpes simplex) of either ear.
11. Dermatitis of the infected ear such as psoriasis or seborrhea that would complicate evaluations.
12. Significant underlying disease such as diabetes, HIV or other immunocompromised conditions or receiving therapy that may cause patient to be immunocompromised.
13. Significant history or current evidence of chronic infectious disease, system disorder, organ disorder or other medical condition that in the Investigator's opinion would place the study patient at undue risk by participation or could jeopardize the integrity of the study evaluations.
14. Investigator believes that severity of infection is such that systemic antibiotics would be the preferred treatment option.
15. Use of any systemic antibacterial products or topical antibacterial products in the ear(s) within 28 days of screening for the study.
16. Use of any systemic anti-inflammatory products or topical anti-inflammatory products in the ear(s) (such as corticosteroids and NSAIDs) within 7 days of screening for the study.
17. Use of any topical or otic medication in the affected ear within 2 weeks prior to screening.
18. Use of any astringents such as vinegar, alcohol or medicated cleansing or swabbing of the ear within 48 hours of the baseline bacterial culture swab.
19. Any known hypersensitivity to ciprofloxacin or other carboxyquinolone derivatives, dexamethasone or corticosteroids or other ingredients of the formulation.
20. Receipt of any drug or device as part of a research study within 30 days prior to dosing.
21. Previous participation in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2013-07; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Clinical Success | Day 14-21
  Evaluation of the difference between the proportions of patients considered a clinical success at the End of Study visit

SECONDARY OUTCOMES:
Resolution of Symptoms | Day 14-21
  The time to complete resolution of disease specific clinically meaningful signs and symptoms at enrollment and the absence of new symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Chandra S Vattikonda, Ph.D., Study Director — Par Pharamceutical, Inc.
Locations (32):
- United States (27):
  - James Donivan Gordon, MD, Tucson, Arizona
  - Nea Baptist Clinic, Jonesboro, Arkansas
  - Applied Reserch Center, Little Rock, Arkansas
  - John Champlin, MD, Carmichael, California
  - Aliance Research, Long Beach, California
  - ENT of South Florida, Boyton Beach, Florida
  - Moore Clinical Research Inc, Fort Myers, Florida
  - Jorge Diaz, MD, Hialeah, Florida
  - San Marcus Research Clinic, Miami, Florida
  - The Medical Consulting Center, Miami, Florida
  - Ormond Medical Arts Pharmaceutical Research Center, Ormond Beach, Florida
  - Winter Park Clinical Research, Winter Park, Florida
  - Research Integrity, LLC, Owensboro, Kentucky
  - Pioneer Clinical Research, Bellevue, Nebraska
  - PMG Research of Raleigh, Raleigh, North Carolina
  - PMG Research of Salisbury, Salisbury, North Carolina
  - Julia Mullen, MD, Cincinnati, Ohio
  - Integrated Medical Research PC, Ashland, Oregon
  - Cyn3rgy, Gresham, Oregon
  - Peak Research LLC, Upper Saint Clair, Pennsylvania
  - John Ansley, MD, Orangeburg, South Carolina
  - Spartanburg and Geer ENT, Spartanburg, South Carolina
  - Monica Davis, MD, Brentwood, Tennessee
  - Gilbert Ledesma, MD, Arlington, Texas
  - West Houston Clinical Research Service, Houston, Texas
  - R-D Clinical Research, Lake Jackson, Texas
  - The Education and Research Foundation Inc., Lynchburg, Virginia
- Puerto Rico (5):
  - SMO The Clinical Research Group, Canovanas, PR
  - Clinical Research Puerto Rico Guayama, Levittown, PR
  - SMO The Clinical Research Group, Naranjito, PR
  - SMO The Clinical Research Group, San Juan, PR
  - SMO The Clinical Resarch Group, Santa Isabel, PR